CLINICAL TRIAL: NCT04235387
Title: Analysis of Haemodynamic Parameters of Patients Undergoing Robotic Prostatectomy
Brief Title: Haemodynamic Changes During Robotic Prostatectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Czech Technical University in Prague (Other)
Collaborators: University Hospital, Motol (Other)
Responsible Party: Sponsor
Other Study IDs: VentRes-2019-03-MR
Record Dates: First submitted 2020-01-13; First posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Robotic Surgical Procedures
Keywords: robotic surgical procedures; laparoscopic surgical procedures; prostatectomy; haemodynamic changes; ventilatory changes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Robotic prostatectomy: All patients undergoing robotic assisted prostatectomy in University Hospital in Motol during the project period. Monitored using standard non-invasive monitoring.
- Laparoscopic prostatectomy: All patients undergoing standard laparoscopic prostatectomy in University Hospital in Motol during the project period. Monitored using standard non-invasive monitoring.

SUMMARY:
The aim of the study is to analyse the haemodynamic and ventilatory changes in patients undergoing robotic prostatectomy, compared to standard laparoscopic prostatectomy.

DETAILED DESCRIPTION:
Prostatectomy is a standard operation, increasingly performed using robotic assistance. During robotic assisted procedures, the intraabdominal pressures are usually higher than in standard laparoscopic operations which can pose a risk of cardiovascular and respiratory adverse effects. The aim of this study is to investigate the haemodynamic and ventilatory effects of robotic assisted prostatectomy, compared to standard laparoscopic prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing prostatectomy in University Hospital in Motol between 1st December 2019 and 30th April 2020

Exclusion Criteria:

* body mass index over 35
* regular use of beta-blocking drugs

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostatectomy performed only in male patients.
Study Population: All patients undergoing prostatectomy in University Hospital in Motol between 1st December 2019 and 30th April 2020.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Haemodynamic changes | Through study completion, an average of 1 year
  Changes in mean arterial pressure.
Ventilatory changes | Through study completion, an average of 1 year
  Changes in peak airway pressure and mean airway pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Vymazal, Ass.prof., Study Chair — University Hospital in Motol
Locations (2):
- Czechia (2):
  - Motol University Hospital, Prague
  - Czech Technical University, Prague